CLINICAL TRIAL: NCT03418207
Title: The Study on the Spatial Distribution of Prostate Cancer by Modified Trans-perineal Template-guided Mapping Biopsy
Brief Title: The Accuracy of Modified TTMB in the Spatial Distribution of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Principal Investigator, Xuefei Ding,MD, Chief physician of urology, Subei People's Hospital of Jiangsu Province
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SubeiPHJP
Record Dates: First submitted 2018-01-23; First posted 2018-02-01 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: TPS system; trans-perineal template-guided mapping biopsy; prostate cancer; spatial distribution; large tissue slice
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTMB for patients (Other): give trans-perineal template-guided mapping biopsy for participants suspected prostate cancer
  Interventions: Procedure: trans-perineal template-guided mapping biopsy

INTERVENTIONS:
Procedure: trans-perineal template-guided mapping biopsy — new super saturation of prostate biopsy technique

SUMMARY:
Investigators plan to use modified TTMB technology to puncture prostate of participants suspected prostate cancer, especially those with the first negative biopsy , but having a rising PSA.Then, Investigators will simulate the spatial distribution of prostate cancer in patients with positive biopsy before radical prostatectomy by way of the TPS software system . And after the radical prostatectomy ,Investigators will simulate the spatial distribution with the help of large tissue slice technique to compare with preoperative simulation ,which to verify the two simulations are consistent.

DETAILED DESCRIPTION:
Investigators mainly plan to determine the accuracy of the modified TTMB technology in combination with the TPS system on the location of the tumor space distribution by comparing the two simulation, which is significant for the accurate focal thearpy.

ELIGIBILITY:
Inclusion Criteria:

1.Male patients;

2.18 yrs and older, and 90 yrs and younger;

3.Rectal examination reveal prostate nodules;

4.B ultrasound, CT or MRI find abnormal images;

5.PSA>4ng/ml, abnormal f/t ratio and PSAD

Exclusion Criteria:

1. Abnormal coagulation function;
2. Severe urinary tract infection;
3. Serious cardiovascular and cerebrovascular disease

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
the spatial distribution based on the biopsy tissue | 2 years
  to simulate the spatial distribution of cancer based on the biopsy tissue contained cancer with the help of TPS system

SECONDARY OUTCOMES:
the spatial distribution based on the large tissue slice technique | 2 years
  to simulate the spatial distribution based on the large tissue slice technique after radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Ding, MD, Principal Investigator — Subei People's Hospital of Jiangsu Province
Locations (1):
- Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran M, Thompson J, Bohm M, Pulbrook M, Moses D, Shnier R, Brenner P, Delprado W, Haynes AM, Savdie R, Stricker PD. Combination of multiparametric MRI and transperineal template-guided mapping biopsy of the prostate to identify candidates for hemi-ablative focal therapy. BJU Int. 2016 Jan;117(1):48-54. doi: 10.1111/bju.13090. Epub 2015 May 11. PMID 25682968